CLINICAL TRIAL: NCT01241253
Title: Glycemic Response of Bean-and-rice Meals in Persons With Type 2 Diabetes Mellitus
Brief Title: Glycemic Response of Bean-and-rice Meals in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: United States Dry Bean Council (Other)
Responsible Party: Principal Investigator, Donna M. Winham, DrPH, Outside Consultant, Arizona State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NTS0020
Record Dates: First submitted 2010-10-27; First posted 2010-11-16 (Estimated); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Blood Glucose; Type 2 Diabetes Mellitus
Keywords: legumes; glycemic response; glucose; type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cross-over study (No Intervention): beans and rice in a 50 gram carbohydrate dose
  Interventions: Other: Whole cooked beans with rice meals

INTERVENTIONS:
Other: Whole cooked beans with rice meals — Three types of bean-and-rice meals all equal to 50 grams available CHO. Control treatment was 50 grams available CHO in the form of white rice alone.
  Other Names: Bush Brothers & Company brand canned beans

SUMMARY:
The study uses a randomized, placebo-controlled experimental design consisting of 4 different test treatments matched on carbohydrate (CHO) content. The three beans are similar in their CHO content amount for ½ cup at ~20 grams CHO. Each of the bean varieties will be served in a ~½ cup serving size with ~ ½ cup of plain steamed white rice (30 grams CHO) for a total of 50 grams of CHO per meal for each of the three test treatments. The 4th placebo or control treatment consists of ~ 7/8 cup of rice alone, an amount consistent with the CHO content of the test meals. Most diabetic meal plans recommend no more than 45-60 grams of CHO per meal. Fifty grams of CHO is a standard amount for glycemic response testing in general.

The investigators hypotheses were:

* The test meals containing the three bean types in combination with white rice will decrease the participants' glycemic response when eaten as part of a meal.
* The reduction in post-prandial glycemia will not differ between bean types in the elicited responses among individuals with type 2 diabetes.

DETAILED DESCRIPTION:
The 4 test treatments will be administered randomly on a different morning, at least one week apart. Participants will be required to consume the entire test treatment meal in 7 minutes while being observed. All test foods will be purchased from local markets. Capillary blood samples will be collected (~50µl) at time 0 (fasting) and at 30, 60, 90, 120 and 180 minutes post-treatment (timing of the post-treatment blood draws started at time 0 [post-treatment], which is when the participant finishes consuming the treatment meal). Venous blood draws for insulin assessment will also be acquired at fasting and then every hour for the three hour study period. Anthropometric measures such as weight, height and waist circumference will be collected at screening and at the start of each test day. Thirteen hours before testing, participants will eat a control meal to reduce variation in glycemic responses on test days due to varying dietary intakes. This control meal will be selected by each participant before the start of the study. They will be provided a gift card to the chain restaurant to use to purchase their own meal. Since subjects serve as their own controls, the meals must be identical before each test draw. Participants will complete 24 hour recall food records the morning of each test day to provide information related to dietary protocol compliance.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects will be between the ages of 35 and 75, have a body mass index value (BMI) between 22-40 kg/m2, be physician diagnosed with type 2 diabetes for at least six (6) months and currently controlling their blood glucose levels using dietary methods, exercise and/or through the use of oral hypoglycemic agents such as Metformin for at least three(3)months, and have an HbA1c <10%.

Exclusion Criteria:

* Exclusion criteria included: the presence of unresolved health issues (e.g. hypertension not controlled by medication), evidence of condition(s) that would influence the participant's ability to complete the study such as gastrointestinal disease, weight changes of ≥10% of the participants body weight within a 6 month period, women who are either pregnant or breastfeeding, allergy to beans or latex, an HbA1c level >10% at screening, and the inability to follow study protocol.

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2009-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Net blood glucose changes over time | fasting baseline glucose at time 0, then 30, 60, 90, 120, 150, and 180 minutes postprandial
  Capillary blood samples were collected via fingerstick using Safe-T-Fill® Lithium Heparin Mini Capillary Collection 125µl tubes (RAM Scientific, Yonkers, NY). Whole blood samples were analyzed for glucose content using the Yellow Springs Instrument Stat Plus Analyzer (YSI Life Sciences, Yellow Springs, OH) immediately after blood collection.

CONTACTS AND LOCATIONS:
Overall Officials: Donna M Winham, DrPH, Principal Investigator — Arizona State University
Locations (1):
- Arizona State University, Nutrition Program, Mesa, Arizona, United States

REFERENCES:
- [Result] Thompson SV, Winham DM, Hutchins AM. Bean and rice meals reduce postprandial glycemic response in adults with type 2 diabetes: a cross-over study. Nutr J. 2012 Apr 11;11:23. doi: 10.1186/1475-2891-11-23. PMID 22494488
- [Result] Hutchins AM, Winham DM, Thompson SV. Phaseolus beans: impact on glycaemic response and chronic disease risk in human subjects. Br J Nutr. 2012 Aug;108 Suppl 1:S52-65. doi: 10.1017/S0007114512000761. PMID 22916816
- [Result] Winham DM, Hutchins AM, Thompson SV. Glycemic Response to Black Beans and Chickpeas as Part of a Rice Meal: A Randomized Cross-Over Trial. Nutrients. 2017 Oct 4;9(10):1095. doi: 10.3390/nu9101095. PMID 28976933